CLINICAL TRIAL: NCT02094703
Title: The Efficacy of Solifenacin Succinate as Adjuvant Therapy for Symptomatic Non-complicated Urinary Tract Infection in Females
Brief Title: The Efficacy of Solifenacin Succinate as Adjuvant Therapy for Urinary Tract Infection in Females
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Collaborators: Astellas Pharma Indonesia Inc. (Industry); Pharos Life Corporation (Industry)
Responsible Party: Principal Investigator, Harrina Erlianti Rahardjo,MD,PhD, MD, PhD, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: URO-SOL-01-2012
Record Dates: First submitted 2014-03-10; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Urinary Tract Infection
Keywords: female; age 18-65 years; storage symptoms; clinical urinary tract infection; non complicated
MeSH Terms: conditions — Urinary Tract Infections | interventions — Levofloxacin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- levofloxacin and solifenacin succinate (Experimental): Levofloxacin 500 mg tablet and solifenacin succinate 5 mg tablet by mouth once daily for 3 days
  Interventions: Drug: Levofloxacin; Drug: Solifenacin succinate
- levofloxacin and placebo (Active Comparator): Levofloxacin 500 mg tablet and placebo (for solifenacin succinate) by mouth once daily for 3 days
  Interventions: Drug: Levofloxacin; Drug: Placebo (for Solifenacin succinate)

INTERVENTIONS:
Drug: Levofloxacin
  Other Names: neslav
Drug: Solifenacin succinate
  Arms: levofloxacin and solifenacin succinate
Drug: Placebo (for Solifenacin succinate)
  Arms: levofloxacin and placebo

SUMMARY:
The efficacy of Solifenacin Succinate 5 mg as adjuvant therapy and levofloxacin (500 mg) for short-term treatment to reduce symptoms in patients with symptomatic non complicated urinary tract infection in females.

ELIGIBILITY:
Inclusion Criteria:

* females (18-65 years old)
* dysuria in symptomatic non complicated urinary tract infection

Exclusion Criteria:

* Pediatric Patients (< 18 years old)
* geriatric Patients (> 65 years old)
* pregnant Patients
* Patients with complicated urinary tract infection
* sexually transmitted infections
* Patients with pathological abnormalities in the urinary bladder, including stone/mass
* Catheter-mounted
* Neurological diseases/disorders
* patients with allergy/hypersensitivity with Levofloxacin/Solifenacin

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with storage symptoms | up to three days

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Jakarta Special Capital Region, Indonesia